CLINICAL TRIAL: NCT04070963
Title: Incidence of Undiagnosed and Poorly Controlled Diabetes Mellitus Among Surgical Patients and Its Association With Perioperative Outcomes: a Single-centre Prospective Cohort Study
Brief Title: Incidence of Poorly Controlled Diabetes in Surgical Population
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201812-00075 C
Record Dates: First submitted 2019-07-28; First posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Diabetes Mellitus
Keywords: Incidence of Diabetes Mellitus; HbA1C
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort: We propose a prospective, observational single-centre pilot study in the PAC (SGH), on participants aged 21 years and above. A HbA1c test will be added to their routine preoperative blood tests. The incidence of newly-diagnosed DM/pre-diabetes (HbA1c ≥6.1%) and poorly controlled DM (HbA1c ≥ 8%), demographic details and presence of significant comorbidities will be analysed.
  Interventions: Other: HbA1C

INTERVENTIONS:
Other: HbA1C — To take additional blood test of HbA1C once patient consented to the study

SUMMARY:
Our study aims to determine the incidence of undiagnosed and poorly controlled diabetes among surgical patients in Singapore using preoperative HbA1c as a screening tool.

DETAILED DESCRIPTION:
The study aims to determine the incidence of undiagnosed and poorly controlled diabetes among surgical patients in Singapore using preoperative HbA1c as a screening tool.

The investigators aim to follow up on the incidence of perioperative complications in this cohort. In the longer term, the investigators hope to evaluate the role of a preoperative diabetic screening and intervention program as an opportunistic "teachable moment" for surgical patients. This may help to achieve greater control of the disease burden in Singapore.

Specific aims:

Specific Aim 1: To establish the incidence of undiagnosed diabetes/prediabetes among surgical patients in Singapore, based on HbA1c level ≥ 6.1% prior to surgery Specific Aim 2: To establish the incidence of poorly-controlled diabetes among surgical patients in Singapore, based on HbA1c level ≥ 8% prior to surgery Specific Aim 3: To identify and characterize any association between preoperative HbA1c level and postoperative outcomes

ELIGIBILITY:
Inclusion Criteria:

1. Age >21 years old
2. able to give informed consent
3. Scheduled to have preoperative blood taken during clinic visit

Exclusion Criteria:

1. Age < 21 years old
2. unable to given informed consent
3. Not required to have routine preoperative blood tests taken

Ages: 21 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients who comes through the pre operative anesthesia clinic due to scheduled elective operation, who fits the inclusion criteria of the study.
Sampling Method: Probability Sample
Enrollment: 888 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-09-01 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Diabetes incidence | 12 months
  To determine the incidence of undiagnosed and poorly controlled diabetes among surgical patients in Singapore

SECONDARY OUTCOMES:
Association of HbA1C levels with post operative complications | 12 months
  To identify and characterize any association between preoperative HbA1c level and postoperative complications, including morbidity and mortality.

CONTACTS AND LOCATIONS:
Locations (1):
- Lim Wan Yen, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Phan TP, Alkema L, Tai ES, Tan KH, Yang Q, Lim WY, Teo YY, Cheng CY, Wang X, Wong TY, Chia KS, Cook AR. Forecasting the burden of type 2 diabetes in Singapore using a demographic epidemiological model of Singapore. BMJ Open Diabetes Res Care. 2014 Jun 11;2(1):e000012. doi: 10.1136/bmjdrc-2013-000012. eCollection 2014. PMID 25452860
- [Background] Wee HL, Ho HK, Li SC. Public awareness of diabetes mellitus in Singapore. Singapore Med J. 2002 Mar;43(3):128-34. PMID 12005338
- [Result] Pang PY, Lim YP, Ong KK, Chua YL, Sin YK. 2015 Young Surgeon's Award Winner: Long-term Prognosis in Patients with Diabetes Mellitus after Coronary Artery Bypass Grafting: A Propensity-Matched Study. Ann Acad Med Singap. 2016 Mar;45(3):83-90. PMID 27146460